CLINICAL TRIAL: NCT01160770
Title: Safety and Effectiveness of Open-Label Clobazam in Subjects With Lennox-Gastaut Syndrome
Acronym: LGS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13109A; OV1004 (Other: Lundbeck LLC ((Formerly Lundbeck Inc. and before that Ovation Pharmaceuticals (OV)))
Record Dates: First submitted 2010-06-18; First posted 2010-07-12 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-02

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Lennox-Gastaut Syndrome (LGS); Epilepsy; Drop Seizures; Clobazam
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsy; Syncope | interventions — Clobazam; Sodium Fluoride; psyton

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clobazam (Experimental)
  Interventions: Drug: Clobazam

INTERVENTIONS:
Drug: Clobazam — Clobazam will be provided in 5 mg, 10 mg and 20 mg tablets and will be dispensed in bottles as needed at each visit. Bottles may be dispensed between visits if necessary. Subjects will start at a common dose level of 0.5 mg/kg, not to exceed 40 mg/day, and must maintain the dose level for 48 hours. After the first 48 hours of the treatment period, investigators will be able to increase, decrease or maintain the subject's dose, up to an approximate maximum daily dose of 2.0 mg/kg (maximum dose of 80 mg/day).
  Other Names: Aedon, Antacastill, Castilium, Clarmyl, Frisium, Karidium, Mefrilan, Mystan, Noiafren, Onfi, Psiton, Psyton, Sentil, Seryl, Urbadan, Urbanil, Urbanol, Urbanyl.

SUMMARY:
The objective of this study is to evaluate the long-term safety and effectiveness of open-label clobazam in the treatment of drop seizures in subjects with LGS.

DETAILED DESCRIPTION:
This multi-center, open-label study is designed to evaluate the long-term safety and effectiveness of clobazam as adjunctive therapy in subjects with LGS. Subjects enrolled in Lundbeck LLC (formerly Ovation Pharmaceuticals, Inc.) sponsored studies 13108A/OV1002/NCT00162981 and 13110A/OV1012/NCT00518713 who either completed the study or who prematurely discontinued were offered the opportunity to rollover into this open-label study. Subjects will start at a common dose level of 0.5 mg/kg, not to exceed 40 mg/day, and must maintain the dose level for 48 hours. After 48 hours, investigators will be able to increase, decrease or maintain the subject's dose, up to a maximum target daily dose of 2.0 mg/kg (maximum dose of 80 mg/day). During the treatment period, seizures will be recorded during the week preceding each study visit or 30 days immediately following each study visit (dependent on Amendment approval). The subject or subject's caregiver will record daily counts of seizures, including drop seizures in the subject's seizure diary.

ELIGIBILITY:
Inclusion Criteria:

* The subject or subject's legally authorized representative (LAR) must sign and date the institutional review board (IRB)/independent ethics committee (IEC) approved Informed Consent Form/Health Insurance Portability and Accountability Act (HIPAA) Authorization (if required) prior to study participation.
* Previous participation in Lundbeck-sponsored LGS study.
* Subject must weigh ≥12.5 kilograms.
* Male or female subjects must have been between 2 and 60 years of age at the time of the enrollment in the Phase 3 double-blind study (13110A/OV1012/NCT00518713) or between 2 and 30 years of age at the time of the enrollment in the Phase 2 double-blind study (13108A/OV1002/NCT00162981) study.
* If female:

  * Subject is either not of childbearing potential, defined as premenarchal, postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or if of childbearing potential, must comply with a method of birth control acceptable to the investigator during the study, for at least 4 weeks prior to study entry and for 4 weeks following completion of the study.
  * Subject is not breastfeeding.
  * Subjects of childbearing potential must have a negative serum pregnancy test at Study Day 1.
* In the investigator's opinion, parent or caregiver must be able to keep an accurate seizure diary.

Exclusion Criteria:

* Greater than 14 days have elapsed since the subject received his/her last dose of study medication in the previous Lundbeck-sponsored LGS study.
* Subject had a serious or severe adverse event in the previous Lundbeck-sponsored LGS study that in the opinion of the investigator was probably or definitely related to clobazam use and precludes safe use of clobazam.
* Subject has had an anoxic episode requiring resuscitation within 6 months of study entry.
* Subject has a history of an allergic reaction or significant sensitivity to benzodiazepines or to any of the other ingredients in clobazam tablets.
* Subject is taking more than 3 concurrent anti-epileptic drugs (AEDs). NOTE: Vagal Nerve Stimulator (VNS) or ketogenic diet is allowed and will not be counted in the three allowed AEDs.
* Subject is currently taking long-term systemic steroids (excluding inhaled medication for asthma treatment) or any other daily medication known to exacerbate epilepsy. An exception will be made of prophylactic medication, for example, for idiopathic nephrotic syndrome or asthma.
* If the subject is taking felbamate, has been taking it for less than 1 year prior to study entry or previous treatment with felbamate resulted in withdrawal due to liver or bone marrow adverse events.
* Subject has experienced an idiosyncratic reaction to an AED, e.g., carbamazepine with resulting aplastic anemia or agranulocytosis, topiramate with resulting metabolic acidosis, felbamate with resulting aplastic anemia or hepatic failure, or lamotrigine with resulting skin irritation and/or rash.
* Subject has shown any clinically significant history of hyper-sensitivity to central nervous system (CNS) active medications leading to neurobehavioral aberrations (e.g., increased biting, scratching, kicking, or hitting).
* Subject has taken or used any investigational drug or device in the 30 days prior to screening, with the exception of clobazam in a Lundbeck-sponsored study.
* Subject has a clinically significant unstable hepatic, hematological, renal, cardiovascular, gastrointestinal, or pulmonary disease or ongoing malignancy.
* Subject has a diagnosis of sleep apnea.
* Subject has a compromised respiratory function or severe respiratory insufficiency.
* Subject has a history of severe muscle weakness, including myasthenia gravis.
* Subject has a clinically significant abnormal laboratory value or electrocardiogram (ECG) abnormality.
* Subject has progressive lesion confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) scan.
* Subject has a history of drug or alcohol abuse.
* Subject has a history of poor compliance on past antiepileptic therapy.
* Subject has inadequate supervision by parent or guardian.
* For any reason, the subject is considered by the investigator to be an unsuitable candidate for the study.

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 267 (Actual)
Dates: Start 2005-12; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Ng YT, Conry J, Paolicchi J, Kernitsky L, Mitchell W, Drummond R, Isojarvi J, Lee D, Owen R; OV-1004 study investigators. Long-term safety and efficacy of clobazam for Lennox-Gastaut syndrome: interim results of an open-label extension study. Epilepsy Behav. 2012 Dec;25(4):687-94. doi: 10.1016/j.yebeh.2012.09.039. Epub 2012 Nov 7. PMID 23141144
- [Result] Ng YT, Conry J, Kernitsky L, Mitchell W, Veidemanis R, Drummond R, Muniz R, Isojarvi J, Lee D, Paolicchi J. Long-Term Safety and Efficacy of Clobazam for Lennox-Gastaut Syndrome: Final Results of an Open-Label Extension Study. Late-Breaking Abstract #1.363 presented at the 66th annual meeting of the American Epilepsy Society, Nov. 30-Dec. 4, 2012, San Diego, California.
- [Derived] Gidal BE, Wechsler RT, Sankar R, Montouris GD, White HS, Cloyd JC, Kane MC, Peng G, Tworek DM, Shen V, Isojarvi J. Deconstructing tolerance with clobazam: Post hoc analyses from an open-label extension study. Neurology. 2016 Oct 25;87(17):1806-1812. doi: 10.1212/WNL.0000000000003253. Epub 2016 Sep 28. PMID 27683846

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled in the LGS studies 13108A/OV1002/NCT00162981 or 13110A/OV1012/NCT00518713 sponsored by Lundbeck LLC who either completed the study or who prematurely discontinued will have the opportunity to rollover into this open-label study.
Groups:
- Clobazam: Start dose was 0.5 mg/kg with a maximum of 40 mg/day to be adjusted; administered as tablets twice daily
Period: Overall Study
Arm/Group | Clobazam
Started | 267
Completed | 188
Not Completed | 79
Not completed — Adverse Event | 10
Not completed — Protocol Violation | 2
Not completed — Subject/parent/caregiver request | 33
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 7
Not completed — Study termination or sponsor request | 1
Not completed — Death | 9
Not completed — Lack of Efficacy | 15
Not completed — Other Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clobazam
Number analyzed (Participants) | 267
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (7.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 163

OUTCOME MEASURES:

1. Primary Outcome: Median Percent Reduction in Average Weekly Rate of Drop Seizures Based on the 7-day Assessment
Description: Number of drop seizures was obtained from seizure diaries
Time Frame: Baseline to month 36
Measure: Median (Full Range); unit: percentage of drop seizures
Arm/Group | Clobazam
Number analyzed (Participants) | 113
percentage of drop seizures | 92.3 [-588 to 100]

2. Primary Outcome: Median Percent Reduction in Average Weekly Rate of Drop Seizures Based on the Last 30-day Assessment
Description: Number of drop seizures was obtained from seizure diaries
Time Frame: Baseline to month 36
Measure: Median (Full Range); unit: percentage of drop seizures
Arm/Group | Clobazam
Number analyzed (Participants) | 121
percentage of drop seizures | 92.7 [-752 to 100]

3. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a ≥25%, ≥50%, ≥75%, 100% Reduction in Drop Seizures Based on the 7-day Assessment
Description: Number of drop seizures obtained from seizure diaries
Time Frame: Baseline to month 36
Measure: Number; unit: percentage of participants
Arm/Group | Clobazam
Number analyzed (Participants) | 113
percentage of participants
  Any reduction | 85.8
  ≥25% reduction | 82.3
  ≥50% reduction | 77.9
  ≥75% reduction | 64.6
  100% reduction | 38.1

4. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a ≥25%, ≥50%, ≥75%, 100% Reduction in Drop Seizures Based on the Last 30-day Assessment
Description: Number of drop seizures obtained from seizure diaries
Time Frame: Baseline to month 36
Measure: Number; unit: percentage of participants
Arm/Group | Clobazam
Number analyzed (Participants) | 121
percentage of participants
  Any reduction | 86.0
  ≥25% reduction | 83.5
  ≥50% reduction | 79.3
  ≥75% reduction | 64.5
  100% reduction | 31.4

5. Secondary Outcome: Investigator Global Evaluations of the Patient's Overall Change in Symptoms
Description: The physician was asked to rate the patient's overall change in symptoms since the beginning of clobazam treatment by checking "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse".
Time Frame: Baseline to month 36
Measure: Number; unit: percentage of participants
Arm/Group | Clobazam
Number analyzed (Participants) | 137
percentage of participants
  VERY MUCH IMPROVED | 35.0
  MUCH IMPROVED | 45.3
  MINIMALLY IMPROVED | 14.6
  NO CHANGE | 2.2
  MINIMALLY WORSE | 0.7
  MUCH WORSE | 1.5
  VERY MUCH WORSE | 0.7

6. Secondary Outcome: Parent/Caregiver Global Evaluations of the Patient's Overall Change in Symptoms
Description: The parent/caregiver was asked to rate the patient's overall change in symptoms since the beginning of clobazam treatment by checking "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse".
Time Frame: Baseline to month 36
Measure: Number; unit: percentage of participants
Arm/Group | Clobazam
Number analyzed (Participants) | 137
percentage of participants
  VERY MUCH IMPROVED | 45.3
  MUCH IMPROVED | 35.0
  MINIMALLY IMPROVED | 11.7
  NO CHANGE | 3.6
  MINIMALLY WORSE | 1.5
  MUCH WORSE | 2.9
  VERY MUCH WORSE | 0.0

ADVERSE EVENTS:
Time Frame: The protocol was written to go up to 60 months treatment however a percentage of patients went beyond 60 months until study completion when commercial product was made available.
Arm/Group | Clobazam
Serious Adverse Events (participants affected / at risk) | 115/267
Other Adverse Events (participants affected / at risk) | 241/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clobazam (N=267)
Anaemia (Blood and lymphatic system disorders) | 4
Anaemia Macrocytic (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Cardio-Respiratory Arrest (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hip Dysplasia (Congenital, familial and genetic disorders) | 1
Talipes (Congenital, familial and genetic disorders) | 2
Hypothalamo-Pituitary Disorder (Endocrine disorders) | 1
Eye Disorder (Eye disorders) | 1
Barrett's Oesophagus (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal Perforation (Gastrointestinal disorders) | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Hiatus Hernia (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 1
Intestinal Obstruction (Gastrointestinal disorders) | 1
Pancreatic Pseudocyst (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Death (General disorders) | 2
Drug Interaction (General disorders) | 1
Oedema Peripheral (General disorders) | 1
Pitting Oedema (General disorders) | 1
Pneumatosis (General disorders) | 1
Pyrexia (General disorders) | 5
Cholecystitis Chronic (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Bronchopneumonia (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 4
Chest Wall Abscess (Infections and infestations) | 1
Clostridium Difficile Colitis (Infections and infestations) | 1
Cystitis Klebsiella (Infections and infestations) | 1
Dengue Fever (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1
Febrile Infection (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Gastroenteritis Viral (Infections and infestations) | 3
Implant Site Infection (Infections and infestations) | 2
Incision Site Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Lobar Pneumonia (Infections and infestations) | 5
Lower Respiratory Tract Infection (Infections and infestations) | 1
Lung Infection Pseudomonal (Infections and infestations) | 2
Oesophageal Candidiasis (Infections and infestations) | 1
Oral Candidiasis (Infections and infestations) | 2
Otitis Media (Infections and infestations) | 2
Periorbital Cellulitis (Infections and infestations) | 1
Peritonsillar Abscess (Infections and infestations) | 1
Pharyngotonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 26
Pneumonia Influenzal (Infections and infestations) | 1
Pneumonia Mycoplasmal (Infections and infestations) | 1
Pneumonia Viral (Infections and infestations) | 2
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1
Respiratory Syncytial Virus Infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 5
Septic Shock (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Staphylococcal Infection (Infections and infestations) | 1
Tooth Abscess (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2
Urinary Tract Infection (Infections and infestations) | 8
Urinary Tract Infection Fungal (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 3
Viral Tracheitis (Infections and infestations) | 2
Bloody Airway Discharge (Injury, poisoning and procedural complications) | 1
Device Malfunction (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Feeding Tube Complication (Injury, poisoning and procedural complications) | 2
Femur Fracture (Injury, poisoning and procedural complications) | 3
Foreign Body Trauma (Injury, poisoning and procedural complications) | 1
Jaw Fracture (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 2
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1
Shunt Malfunction (Injury, poisoning and procedural complications) | 2
Therapeutic Agent Toxicity (Injury, poisoning and procedural complications) | 5
Ventriculoperitoneal Shunt Malfunction (Injury, poisoning and procedural complications) | 1
Electroencephalogram (Investigations) | 2
Hepatic Enzyme Increased (Investigations) | 1
Oxygen Saturation Decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Failure To Thrive (Metabolism and nutrition disorders) | 1
Feeding Disorder (Metabolism and nutrition disorders) | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophagia (Metabolism and nutrition disorders) | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1
Joint Contracture (Musculoskeletal and connective tissue disorders) | 1
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 2
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 5
Atonic Seizures (Nervous system disorders) | 1
Brain Injury (Nervous system disorders) | 1
Complex Partial Seizures (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 30
Dystonia (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Epilepsy (Nervous system disorders) | 2
Grand Mal Convulsion (Nervous system disorders) | 4
Guillain-Barre Syndrome (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Intracranial Hypotension (Nervous system disorders) | 1
Lennox-Gastaut Syndrome (Nervous system disorders) | 5
Lethargy (Nervous system disorders) | 1
Muscle Spasticity (Nervous system disorders) | 1
Myoclonic Epilepsy (Nervous system disorders) | 1
Petit Mal Epilepsy (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 1
Status Epilepticus (Nervous system disorders) | 11
Tremor (Nervous system disorders) | 1
Abnormal Behaviour (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Mental Status Changes (Psychiatric disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 1
Trigonitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Choking (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Diaphragmatic Hernia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 15
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 4
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 3
Swelling Face (Skin and subcutaneous tissue disorders) | 1
Activities Of Daily Living Impaired (Social circumstances) | 1
Brain Operation (Surgical and medical procedures) | 1
Medical Diet (Surgical and medical procedures) | 1
Spinal Operation (Surgical and medical procedures) | 1
Vagal Nerve Stimulator Implantation (Surgical and medical procedures) | 4
Deep Vein Thrombosis (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Venous Thrombosis Limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clobazam (N=267)
Constipation (Gastrointestinal disorders) | 35
Diarrhoea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 20
Fatigue (General disorders) | 18
Pyrexia (General disorders) | 48
Ear Infection (Infections and infestations) | 15
Gastroenteritis (Infections and infestations) | 14
Influenza (Infections and infestations) | 17
Nasopharyngitis (Infections and infestations) | 31
Otitis Media (Infections and infestations) | 42
Pharyngitis Streptococcal (Infections and infestations) | 18
Pneumonia (Infections and infestations) | 29
Sinusitis (Infections and infestations) | 32
Upper Respiratory Tract Infection (Infections and infestations) | 75
Urinary Tract Infection (Infections and infestations) | 35
Viral Infection (Infections and infestations) | 29
Contusion (Injury, poisoning and procedural complications) | 21
Fall (Injury, poisoning and procedural complications) | 44
Skin Laceration (Injury, poisoning and procedural complications) | 24
Decreased Appetite (Metabolism and nutrition disorders) | 14
Drooling (Nervous system disorders) | 22
Lethargy (Nervous system disorders) | 26
Sedation (Nervous system disorders) | 21
Somnolence (Nervous system disorders) | 45
Aggression (Psychiatric disorders) | 22
Insomnia (Psychiatric disorders) | 31
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review and approve all proposed abstracts, manuscripts, or presentations regarding this study prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.